CLINICAL TRIAL: NCT02936518
Title: Anterior Lingual Frenectomy is Inadequate in Improving Breastfeeding Outcomes: a Prospective Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Oregon Clinic (Other)
Responsible Party: Principal Investigator, Bobak Ghaheri, MD, Otolaryngologist/Head and Neck Surgeon, The Oregon Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOC ENT 2
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Ankyloglossia; Breastfeeding
Keywords: ankyloglossia; breastfeeding; lip tie
MeSH Terms: conditions — Ankyloglossia; Breast Feeding; lip tie

ARMS (1):
- Intervention (Experimental)
  Interventions: Procedure: Lingual frenotomy and/or maxillary labial frenectomy

INTERVENTIONS:
Procedure: Lingual frenotomy and/or maxillary labial frenectomy

SUMMARY:
A previously published study (https://www.ncbi.nlm.nih.gov/pubmed/27641715) identified breastfeeding improvements following lingual frenotomy and/or maxillary labial frenectomy. In the previous cohort, babies were excluded from the study if they had previously undergone an attempted frenotomy prior to seeing the P.I. in the office. The proposed study will only look at those babies who did undergo a previous frenotomy to determine:

1. the presence of continued problematic breastfeeding symptoms
2. if further tongue tie or lip tie release improves those outcomes

ELIGIBILITY:
Inclusion Criteria:

* Healthy babies who are breastfeeding
* Had a previous frenotomy prior to presenting to the P.I.

Exclusion Criteria:

* Twins, triplets
* Maternal breast surgery or IGT
* Premature birth
* Significant heart/lung/brain disease of infant

Ages: 1 Day to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Nipple pain | 1 week post-procedure
Reflux (i-GERQ-R) | 1 week and 1 month post-procedure
Maternal breastfeeding self-efficacy (BSES-SF) | 1 week and 1 month post-procedure

REFERENCES:
- [Background] O'Callahan C, Macary S, Clemente S. The effects of office-based frenotomy for anterior and posterior ankyloglossia on breastfeeding. Int J Pediatr Otorhinolaryngol. 2013 May;77(5):827-32. doi: 10.1016/j.ijporl.2013.02.022. Epub 2013 Mar 22. PMID 23523198
- [Background] Geddes DT, Langton DB, Gollow I, Jacobs LA, Hartmann PE, Simmer K. Frenulotomy for breastfeeding infants with ankyloglossia: effect on milk removal and sucking mechanism as imaged by ultrasound. Pediatrics. 2008 Jul;122(1):e188-94. doi: 10.1542/peds.2007-2553. Epub 2008 Jun 23. PMID 18573859
- [Background] Ghaheri BA, Cole M, Fausel SC, Chuop M, Mace JC. Breastfeeding improvement following tongue-tie and lip-tie release: A prospective cohort study. Laryngoscope. 2017 May;127(5):1217-1223. doi: 10.1002/lary.26306. Epub 2016 Sep 19. PMID 27641715